CLINICAL TRIAL: NCT06514560
Title: OPTImizing MIltefosine Treatment for Cutaneous LEISHmaniasis Patients
Acronym: OPTIMILEISH
Status: Recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Alert Hospital, Ethiopia (Other); Armauer Hansen Research Institute, Ethiopia (Other); Uppsala University (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1708/23
Record Dates: First submitted 2024-06-20; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cutaneous Leishmaniases
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — miltefosine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots for PK analysis Microbiopsy from skin for PCR analysis Routine Skin slit smear for genomic sequencing optional 2mm punch biopsy for PK analysis optional microbiopsy for PK analysis Serum sample for biobanking WB sample for biobanking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-allometric dosing: 40 patients who will not use allometric dosing will be included
  miltefosine will be given based on weight: 30-45 kg: 100mg miltefosine per day >45 kg: 150mg miltefosine per day
  Interventions: Drug: Miltefosine
- allometric dosing (weight below 30 kg): 40 patients who weigh less than 30kg and therefore get allometric dosing will be recruited.
  Dosing is given based on weight, height, and sex, according to Dorlo et al 2012
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — Miltefosine will be prescribed by the treating physician for a minimum of 4 weeks. If treatment response is not sufficient, treatment extension could be decided by the treating physician up to 8 weeks

SUMMARY:
While there are indications that 28 days of miltefosine is not sufficient for treating CL by L. aethiopica, a better understanding of what happens in terms of parasite clearance and drug dosing is lacking. In this study, longitudinal measurements of parasite and drug concentrations during treatment are done to monitor parasite kinetics as well as pharmacokinetics. This data will be crucial to provide more information on duration and dosing of miltefosine in CL patients globally, and in Ethiopia and pediatric patients in particular.

DETAILED DESCRIPTION:
In this project, parasite dynamics and miltefosine pharmacokinetics in the skin and blood during routine durations of miltefosine treatment (4-8 weeks) are studied with the aim to provide evidence to optimize miltefosine dosing for treatment of CL. By also studying these factors in children who get allometric miltefosine dosing, data which can be used to adapt the current allometric dosing scheme specifically to children with CL will be produced. Exploratory objectives will look into searching for more objective outcome assessment measures, resistance, helminth infection and nutritional status as potential factors affecting treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or parasitological (microscopy or PCR) confirmation of leishmaniasis
* Age >2
* Clinical decision to start miltefosine treatment as systemic treatment
* In case of females of child-bearing age: willing to take contraceptive for 6 months (parenteral or IUD or implant)
* Willing and able to provide informed consent
* Willing to be hospitalized for the duration of treatment

Exclusion Criteria:

* Currently on treatment or having received modern treatment for leishmaniasis in the last 3 months
* Pregnant (pregnancy test at D0) or breastfeeding
* Unlikely to come for follow-up visits
* Abnormal lab values Hemoglobin <5.0g/100mL Platelets <50 x 10^9/L White blood count <1 x 10^9/L ASAT/ALAT >3x upper normal range Creatinine above the normal limit

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 40 children on allometric dosing and 40 other patients will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Miltefosine plasma concentrations - Area under the plasma concentration versus time curve (AUC) | Day 0, Day 3, Day 7, Day 14, Day 21, Day 28, Day 42/Day 56, Day 90, Day 180
  Determined by LC-MS/MS, miltefosine pharmacokinetics are assessed through calculation of the area under the plasma concentration-time curve from start of treatment until end of treatment (AUC0-EoT), stratified by whether patients received allometric dosing or not.
Miltefosine plasma concentrations - Maximum plasma concentration (Cmax) | Day 0, Day 3, Day 7, Day 14, Day 21, Day 28, Day 42/Day 56, Day 90, Day 180
  Determined by LC-MS/MS, stratified by whether patients received allometric dosing or not.
MIltefosine plasma concentrations - Time of maximum concentration (Tmax) | Day 0, Day 3, Day 7, Day 14, Day 21, Day 28, Day 42/Day 56, Day 90, Day 180
  Determined by LC-MS/MS, stratified by whether patients received allometric dosing or not.

SECONDARY OUTCOMES:
Parasite kinetics in blood and skin | Day 0, Day 3, Day 7, Day 14, Day 21, Day 28, Day 42/Day 56, Day 90, Day 180
  To determine parasite kinetics in terms of Ct-values in blood and skin (microbiopsy sample) measured by quantitative PCR
Adapted allometric dosing scheme specifically for children with CL | Day 0, Day 3, Day 7, Day 14, Day 21, Day 28, Day 42/Day 56, Day 90, Day 180
  Population PK and PK-PD analysis of the relationship between miltefosine exposure and parasite kinetics will be done at UU, based on results from miltefosine plasma concentrations. Structural pharmacokinetic modelling will be used to develop and simulate alternative dosing schemes for children with CL, using Monte Carlo simulations.
Treatment outcomes of patients on miltefosine treatment | Day 28, day 90 and day 180
  Clinical cure rate determined by complete flattening, complete reepithelization and absence of erythema, crustation, and swelling
Assess safety of miltefosine | Day 28
  Side-effects: number and proportion of patients with adverse events

OTHER OUTCOMES:
To explore optimization of outcome assessment using a 3D scanner | Day 28, Day 90, Day 180
  Machine learning models will be built to explore accuracy (% correctly predicted) of 3D scanning models to predict clinical outcomes.
To explore whether nutritional status in CL patients is related to treatment outcomes | Nutritional status at Day 0, outcome at Day 90/Day 180
  Logistic regression models will be made with clinical cure/no cure as outcome, and nutritional status measured through Z-scores as predictor.
To explore whether helminth infection in CL patients is related to treatment outcomes | Helminth infection at Day 0, outcome at Day 90/Day 180
  Logistic regression models will be made with clinical cure/no cure as outcome, and helminth infection (determined as present/not present by wet mount stool exam) as predictor.
To explore sequencing to detect intrinsic and acquired resistance markers for miltefosine | Day 0, Day 28/Day 42/Day 56, unscheduled visit
  Whole genome sequencing will be done at AHRI to check for intrinsic (before treatment samples) and acquired resistance (relapse and end of treatment samples).
To explore skin tissue miltefosine concentrations | Day 28/Day 42/Day 56
  Measured by LC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Van Henten, Principal Investigator — Institute of Tropical Medicine
Locations (1):
- Africa Leprosy, Tuberculosis, Rehabilitation and Training (ALERT) Hospital, Addis Ababa, Ethiopia